CLINICAL TRIAL: NCT06890026
Title: Durability of Three Monthly Loading Doses With Faricimab Injections in Patients With Treatment-naïve Neovascular Age-related Macular Degeneration
Brief Title: Durability of Three Monthly Loading Doses With Faricimab in Treatment-naïve Neovascular Age-related Macular Degeneration
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: p-2024-16973
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD); Treatment-naïve
Keywords: Neovascular Age-related Macular Degeneration; anti-VEGF; faricimab; loading dose
MeSH Terms: interventions — faricimab; Intravitreal Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Faricimab Injection [Vabysmo] — The procedures were carried out according to the local standard protocol, which involved applying 2-3 drops of topical tetracaine anesthesia, using an eye speculum, disinfecting with 5% povidone-iodine, employing a 33G needle, marking the injection site 3.5 mm posterior to the limbus with calipers in either the superotemporal or inferotemporal quadrant, applying a sterile cotton tip for tamponade after needle removal, and omitting post-procedure antibiotics.
  Other Names: Intravitreal injection

SUMMARY:
Neovascular Age-Related Macular Degeneration (nAMD) is a one of the leading causes of irreversible vision loss among the elderly in developed countries. The implementation of anti-VEGF therapies in the last decades has significantly improved AMD management. Faricimab (Vabysmo®), a bispecific antibody targeting both Vascular Endothelial Growth Factor A (VEGF-A) and Angiopoietin-2 (Ang-2), offers enhanced disease control by both inhibiting angiogenesis and stabilizing blood vessels to prevent inflammation and leakage. Faricimab is thought to potentially reduce the frequency of injections compared to therapies targeting only VEGF-A. A key aspect of evaluating its efficacy is understanding the interval before the need for subsequent injections following the initial loading dose. Treatment with intravitreal anti-VEGF injections would typically start with three injections administered at four-weekly intervals, however faricimab is recommended to be started with four loading injections. Our department routinely initiates anti-VEGF therapy with 3 loading doses and then follows an observe-and-plan regimen. This routine was continued with faricimab injections as well despite the manufacturer's recommendation of 4 monthly loading doses.

Determining the optimal interval for reinjection is crucial for reducing treatment burden and improving patient quality of life.

This study aims to assess the durability of a loading dose of 3 faricimab injections, the need for a follow-up checkup at 4 weeks post-loading and functional outcomes post-loading in treatment-naive patients with neovascular age-related macular degeneration (nAMD),

ELIGIBILITY:
Inclusion criteria

* Age of 50 years or older
* Treatment-naïve patients diagnosed with nAMD who have received a loading dose with intravitreal faricimab
* Follow-up data available until the next subsequent faricimab injection after the loading dose, OR if no injections were indicated following the loading dose, follow-up data for at least 4 months

Exclusion criteria

* History of previous anti-VEGF treatment.
* Neovascular conditions other than AMD (e.g., choroidal neovascularization due to other causes) or co-existence of other retinal disease in the study eye
* Intraocular surgery in the study eye during the loading dose or prior to the first follow-up visit after the loading dose.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Capital Region of Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 828 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Durability of the loadings dose with 3 faricimab injections | 01/NOV/2023 - 31/AUG/2024
  Defined as the time from the third injection in the loading dose series to the next required faricimab injection among those needing reinjection (in weeks).

SECONDARY OUTCOMES:
Proportion of patients with no need for a new injection at the first post-loading dose follow-up visit at 4 weeks. | 01/NOV/2023 - 31/AUG/2024
  Described in percentage
Change in best-corrected visual acuity (BCVA) following the loading phase with faricimab at 4 weeks. | 01/NOV/2023 - 31/AUG/2024
  Described in ETRDS letters

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Schneider, MD, PhD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Department of Ophthalmology, Rigshospitalet, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heier JS, Khanani AM, Quezada Ruiz C, Basu K, Ferrone PJ, Brittain C, Figueroa MS, Lin H, Holz FG, Patel V, Lai TYY, Silverman D, Regillo C, Swaminathan B, Viola F, Cheung CMG, Wong TY; TENAYA and LUCERNE Investigators. Efficacy, durability, and safety of intravitreal faricimab up to every 16 weeks for neovascular age-related macular degeneration (TENAYA and LUCERNE): two randomised, double-masked, phase 3, non-inferiority trials. Lancet. 2022 Feb 19;399(10326):729-740. doi: 10.1016/S0140-6736(22)00010-1. Epub 2022 Jan 24. PMID 35085502
- [Background] Freund KB, Mrejen S, Gallego-Pinazo R. An update on the pharmacotherapy of neovascular age-related macular degeneration. Expert Opin Pharmacother. 2013 Jun;14(8):1017-28. doi: 10.1517/14656566.2013.787410. Epub 2013 Apr 8. PMID 23560774
- [Background] Li JQ, Welchowski T, Schmid M, Mauschitz MM, Holz FG, Finger RP. Prevalence and incidence of age-related macular degeneration in Europe: a systematic review and meta-analysis. Br J Ophthalmol. 2020 Aug;104(8):1077-1084. doi: 10.1136/bjophthalmol-2019-314422. Epub 2019 Nov 11. PMID 31712255